CLINICAL TRIAL: NCT06571708
Title: A Phase 2, Randomized, Open-label Study of Gemcitabine/Cisplatin Plus Cemiplimab (REGN2810, Anti-PD-1) With or Without Fianlimab (REGN3767, Anti-LAG-3) for Organ Preservation in Patients With Localized Muscle-invasive Bladder Cancer (NeoSTOP-IT)
Brief Title: Gemcitabine/Cisplatin Plus Cemiplimab With or Without Fianlimab in Localized Muscle-invasive Bladder Cancer (NeoSTOP-IT)
Acronym: NeoSTOP-IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Alexander Z. Wei, MD, Assistant Professor of Medicine at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAV3927
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma
Keywords: Urothelial Predominant Histology
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Gemcitabine/Cisplatin/Cemiplimab (Experimental): * Gemcitabine 1000 mg/m^2 IV (days 1 and 8 of 21 day for 4 cycles)
  * Cisplatin 70 mg/m^2 IV (day 1 of 21 day cycle for 4 cycles) or renally-dosed split-dose -cisplatin 35 m/m^2 IV (day 1 and 8 of 21 day cycle for 4 cycles)
  * Cemiplimab (REGN 2810) 350 mg IV every 3 weeks (17 cycles)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Cemiplimab
- Group 2: Gemcitabine/Cisplatin/Cemiplimab/Fianlimab (Experimental): * Gemcitabine 1000 mg/m2 IV (days 1 and 8 of 21 day cycle for 4 cycles)
  * Cisplatin 70 mg/m2 IV (day 1 of 21 day cycle for 4 cycles) or renally-dosed split-dose cisplatin 35 m/m2 IV (day 1 and 8 of 21 day cycle for 4 cycles )
  * Cemiplimab (REGN 2810) 350mg IV every 3 weeks (4 cycles)
  * Fianlimab (REGN3767) 1600mg IV every 3 weeks (4 cycles)
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Cemiplimab; Drug: Fianlimab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 IV
Drug: Cisplatin — Cisplatin 70 mg/m^2 IV or renally-dosed split-dose cisplatin 35 m/m^2 IV
Drug: Cemiplimab — Cemiplimab 350mg IV
  Other Names: REGN 2810
Drug: Fianlimab — Fianlimab 1600mg IV
  Other Names: REGN3767
  Arms: Group 2: Gemcitabine/Cisplatin/Cemiplimab/Fianlimab

SUMMARY:
The goal of this clinical trial is to learn if gemcitabine/cisplatin plus cemiplimab with or without fianlimab works to treat bladder cancer in adults. The main question it aims to answer is: Can gemcitabine, cisplatin, and cemiplimab with or without fianlimab treat bladder cancer?

Participants will be randomly selected (like the loss of a coin) to treatment with gemcitabine, cisplatin, cemiplimab, and fianlimab or gemcitabine, cisplatin, and cemiplimab.

Participants will:

* Undergo transurethral resection of bladder tumor (TURBT) followed by the start of treatment, receive 4 cycles of treatment (21 day cycles)
* After 4 cycles of treatment, patients will undergo repeat maximal TURBT with imaging
* Participants with a complete response will continue maintenance cemiplimab or cemiplimab/fianlimab for 13 more cycles with imaging every 3 months
* Participants without a complete clinical response will undergo cystectomy (bladder surgery).

DETAILED DESCRIPTION:
This is a phase 2, open-label, randomized trial with continuous toxicity monitoring to ensure safety using Bayesian toxicity monitoring, which will evaluate treatment with doublet platinum-based chemotherapy (gemcitabine and cisplatin) plus cemiplimab (REGN2810) with or without fianlimab (REGN3767) for localized muscle-invasive bladder cancer (MIBC). Participants will be randomized to 4 cycles of 3 weeks each (12 weeks total) with gemcitabine, cisplatin, and cemiplimab with or without fianlimab. Participants achieving a clinical complete response will continue 13 more cycles of immunotherapy (39 weeks total). The total duration of systemic treatment, including neoadjuvant therapy, will be 52 weeks.

In addition to the actual time on treatment, there will be time off treatment for recovery after neoadjuvant treatment and before adjuvant treatment. First, between the neoadjuvant phase and cystoscopy (with TURBT for residual disease), there will be up to 4 weeks off treatment. In between the cystoscopy/TURBT and start of adjuvant immunotherapy, there will be an additional up to 4 week interval for recovery. Participants will have regularly scheduled study visits at the clinical site on Day 1 and Day 8 of every three-week cycle in the neoadjuvant setting, where continuous assessment, including treatment response and safety assessments, will be performed. These will include laboratory tests, taking of vital signs, and physical examinations. In the adjuvant setting for participants who continue to maintenance immunotherapy, participants will have regularly scheduled study visits at the clinical site on Day 1 of every three-week cycle.

Response to treatment will be determined by three modalities. First, CT scans (chest, abdomen, and pelvis with and without contrast) to ensure no metastatic disease. For participants who are unable to get a CT scan w/ contrast due to renal function (or any other reason), an MRI with and without contrast may be used instead. Scans are required at baseline and every 3 months in the adjuvant setting for participants who continue on with maintenance immunotherapy. Second, all participants will undergo post-treatment cystoscopy every 3 months while on treatment. Third, all participants will undergo post-treatment urine cytology every 3 months while on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on day of signing informed consent.
* Life expectancy > 12 months.
* Performance status of 0-1 using the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Histologically confirmed muscle-invasive urothelial carcinoma of the bladder defined as T2-T3, N0, M0 stage. Mixed histology is permitted if there is a urothelial component. Upper tract disease in not permitted.
* Prior Bacillus Calmette-Guerin (BCG) or other intravesical treatment of non-muscle invasive bladder cancer is permitted if completed at least 6 weeks prior to initiating study treatment. Only one course (includes induction + maintenance) of BCG or intravesical therapy is permitted.
* No metastatic disease based on cross-sectional imaging.
* Considered cisplatin eligible based on protocol specified criteria.
* Not received any adjuvant or neoadjuvant chemotherapy or immunotherapy.
* Agree to pre- and post-treatment TURBT as well as surveillance with cystoscopies, cross-sectional imaging, and urine cytology unless medically contraindicated in the opinion of the treating physician, and discussed with the principal investigator

Exclusion Criteria:

* Concurrent upper urinary tract (i.e., ureter, renal pelvis) invasive urothelial carcinoma. (NOTE: Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post- treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible).
* Received prior immune checkpoint inhibitors (including anti-PD-1, anti-PD-L1, anti-CTLA4, anti-LAG-3 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways ), as well as cellular vaccines, cellular therapies, or systemic oncolytic virus therapy.
* Received bladder-directed radiation therapy previously for bladder cancer.
* Received prior systemic chemotherapy for muscle-invasive bladder cancer.
* Receiving any other investigational agents concurrently or within 4 weeks of start of treatment.
* Had a solid organ or hematologic transplant.
* Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (at a dose greater than 10mg/day of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Has a history of myocarditis.
* Patients with another active second malignancy other than non-melanoma skin cancers.
* Has a known history of, or any evidence of, interstitial lung disease or active noninfectious pneumonitis.
* Has an active infection requiring systemic therapy.
* History or current evidence of significant (Common Terminology Criteria for Adverse Events (CTCAE) grade ≥2) local or systemic infection (eg, cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
* Has a history of current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection.
* Is pregnant or is a breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response | 16 weeks
  Rate of clinical complete response after 4 cycles of neoadjuvant chemoimmunotherapy. Complete clinical response will be defined as:
  * No high-grade malignancy on repeat TURBT
  * No malignant cells on urine cytology
  * No definitive evidence of invasive local or metastatic disease on cross-sectional imaging (CT chest, abdomen, and pelvis with contrast or, if renal dysfunction, MRI with contrast)
  Cytoscopy and imaging should occur within 4 weeks of end of neoadjuvant therapy.

SECONDARY OUTCOMES:
Number of Adverse Events | 30 days after last dose of treatment, up to 56 weeks
  Defined as the occurrence of any adverse event (AE) related to the investigational drugs at any point on treatment until 30 days after the last dose of treatment. AEs as evaluated per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Bladder-intact survival | Up to 5 years
  Bladder-intact survival is defined as the time from start of treatment until cystectomy or death.
Recurrence-free survival | Up to 5 years
  Recurrence-free survival is defined as the time from start of treatment until disease recurrence or death. Recurrence-survival will only be measured in patients who achieve a clinical complete response.
Overall survival | Up to 5 years
  Overall survival is defined as the time from start of treatment until death.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Z Wei, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York, United States